CLINICAL TRIAL: NCT00454974
Title: Preliminary Study to Assess the Safety and Efficacy of a Wearable Artificial Kidney Device for the Treatment of Patients With Endstage Renal Failure
Brief Title: Pilot Study of Wearable Artificial Kidney
Acronym: WAK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royal Free Hampstead NHS Trust (Other)
Collaborators: Xcorporeal (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD7465; R&D Number 7465
Record Dates: First submitted 2007-03-29; First posted 2007-04-02 (Estimated); Last update posted 2007-04-02 (Estimated); Status verified 2007-03

CONDITIONS: Renal Failure
Keywords: end stage renal failure; dialysis; wearable artificial kidney
MeSH Terms: conditions — Renal Insufficiency; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Wearable artificial kidney

SUMMARY:
This is a pilot study of a wearable type of kidney dialysis machine to treat patients with chronic kidney disease.

DETAILED DESCRIPTION:
This is a pilot study to evaluate the clearances, tolerability and safety of a wearable artificial kidney device for treating patients with chronic kidney failure.

ELIGIBILITY:
Inclusion Criteria:

* End stage renal failure
* Regular haemodialysis
* Cardiovascular stability
* Stable vascular access

Exclusion Criteria:

* Allergy to heparin or ethylene oxide
* Recent cardiovascular or neurological event
* Unable to provide informed consent
* Age < 18

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8
Dates: Start 2007-03; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
urea, potassium, phosphate and B2M clearances
safety - cardiovascular,no hemolysis, bleeding, infection
no ammonia generation from sorbents, control of acid base balance

SECONDARY OUTCOMES:
fluid removal
patient satisfaction questionnaire
affect of treatment of cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Victor Gurra, MD, Principal Investigator — Cedars Sinai, Los Angeles, USA
Locations (1):
- UCL Center for Nephrology, London, London, United Kingdom

REFERENCES:
- [Background] Gura V, Beizai M, Ezon C, Polaschegg HD. Continuous renal replacement therapy for end-stage renal disease. The wearable artificial kidney (WAK). Contrib Nephrol. 2005;149:325-333. doi: 10.1159/000085694. PMID 15876856
- [Derived] Gura V, Davenport A, Beizai M, Ezon C, Ronco C. Beta2-microglobulin and phosphate clearances using a wearable artificial kidney: a pilot study. Am J Kidney Dis. 2009 Jul;54(1):104-11. doi: 10.1053/j.ajkd.2009.02.006. Epub 2009 Apr 19. PMID 19376616